CLINICAL TRIAL: NCT03846271
Title: The Effects of Intranasal Oxytocin on Reward Sensitivity and Performance Monitoring During Reinforcement Learning: an ERP Study
Brief Title: Effects of Oxytocin on Reinforcement Learning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-61
Record Dates: First submitted 2019-01-25; First posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Learning Disabilities
Keywords: Oxytocin; performance monitoring; reinforcement learning
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled double-blind within-subject design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin then placebo (Experimental): Participants first receive oxytocin (24 IU). After a washout period of 2 weeks, they receive placebo.
  Interventions: Drug: intranasal oxytocin; Drug: intranasal placebo
- Placebo then oxytocin (Experimental): Participants first receive placebo. After a washout period of 2 weeks, they receive oxytocin (24 IU).
  Interventions: Drug: intranasal oxytocin; Drug: intranasal placebo

INTERVENTIONS:
Drug: intranasal oxytocin — 24 IU of oxytocin nasal spray will be applied to each subject.
Drug: intranasal placebo — an identical amount of placebo nasal spray will be applied to each subject.

SUMMARY:
The main aim of the study is to investigate whether intranasal oxytocin (24IU) influences reward sensitivity and performance monitoring during reinforcement learning.

DETAILED DESCRIPTION:
A double-blind, within-subject, placebo-controlled pharmacological EEG design will be employed. A total of 35 healthy male subjects will be recruited which will receive either intranasal placebo or oxytocin (24IU) on two separate study days (order counter-balanced, washout period at least 2 weeks). 45 minutes after treatment subjects will undergo a probabilistic feedback reinforcement learning paradigm with concurrent EEG acquisition. During the paradigm subjects will learn the reward probabilities of two different visual stimuli from probabilistic feedback provided by social stimuli (positive, negative emoticon). The paradigm includes an initial acquisition phase and a subsequent test phase.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-30
* Male sex
* Right handedness

Exclusion Criteria:

* History of brain injury
* Current or history of psychiatric, neurological or internist disorder
* Current or regular use of medication, psychotropic substances, including nicotine
* Contraindications for Oxytocin

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-12-04 (Actual); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Neural index: Event-related potential: Feedback Related Negativity (FRN) during acquisition phase | 45-105 minutes after treatment administration
  Feedback Related Negativity (FRN): a negative ERP component evoked by negative feedback relative to positive feedback during the acquisition phase will be compared between the oxytocin and placebo treatment conditions.
Neural index: Event-related potential: Error Related Negativity (ERN) during the test phase | 45-105 minutes after treatment administration
  Error Related Negativity (ERN): a negative ERP component evoked by incorrect responses relative to correct responses during the test phase will be compared between the oxytocin and placebo treatment conditions.

SECONDARY OUTCOMES:
Behavioral index: Response accuracy to superior stimuli during the acquisition phase | 45-105 minutes after treatment administration
  Correct responses are defined as choices of the stimulus associated with higher probability positive feedback during the acquisition phase. Effects of treatment will be analyzed by comparing the performance between the two treatment conditions.
Behavioral index: Response accuracy to stimuli associated with highest probability positive feedback during the test phase | 45-105 minutes after treatment administration
  Correct responses are defined as choices of the stimulus associated with highest probability positive feedback as learned in the acquisition phase. Effects of treatment will be analyzed by comparing the performance between the two treatment conditions.
Response accuracy avoiding stimuli associated with highest probability negative feedback in the test phase. | 45-105 minutes after treatment administration
  Correct responses are defined as avoidance choices of stimuli associated with highest probability negative feedback as learned in the acquisition phase. Effects of treatment will be analyzed by comparing the performance between the two treatment conditions.
Response accuracy in response to superior stimuli associated with relative higher probability positive feedback in the test phase. | 45-105 minutes after treatment administration
  Correct responses are defined as choices of the stimulus associated with higher probability positive feedback. Note that stimuli pairs in this measurement are all associated with positive feedback. Effects of treatment will be analyzed by comparing the performance between the two treatment conditions.
Response accuracy avoiding stimuli associated with higher probability negative feedback in the test phase. | 45-105 minutes after treatment administration
  Correct responses are defined as avoidance choices of stimuli associated with higher probability negative feedback. Note that stimuli pairs in this measurement are all associated with negative feedback. Effects of treatment will be analyzed by comparing the performance between the two treatment conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Kendrick, PhD, Principal Investigator — University of Electronic Science and Technology of China(UESTC)
Locations (1):
- University of Electronic Science and Technology of China(UESTC), Chengdu, Sichuan, China